CLINICAL TRIAL: NCT01113632
Title: Phase II Trial of Ofatumumab for Older Patients and Patients Who Refuse Fludarabine-Based Regimens With Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Brief Title: Ofatumumab for Patients With Previously Untreated Chronic Lymphocytic Leukemia or Small Lymphocytic Lymphoma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: SCRI Development Innovations, LLC (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SCRI CLL 11
Record Dates: First submitted 2010-04-28; First posted 2010-04-30 (Estimated); Results first posted 2015-06-04 (Estimated); Last update posted 2016-09-20 (Estimated); Status verified 2016-08

CONDITIONS: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma
Keywords: Chronic Lymphocytic Leukemia; Small Lymphocytic Lymphoma; Ofatumumab
MeSH Terms: conditions — Leukemia, Lymphocytic, Chronic, B-Cell | interventions — ofatumumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Ofatumumab 1000mg (Experimental): Ofatumumab 300mg IV Day 1 followed by ofatumumab 1000mg weekly for a total of 8 weeks
  Interventions: Drug: Ofatumumab
- Ofatumumab 2000mg (Experimental): Ofatumumab 300mg IV Day 1 followed by ofatumumab 2000mg weekly for a total of 8 weeks
  Interventions: Drug: Ofatumumab

INTERVENTIONS:
Drug: Ofatumumab — IV infusion once weekly for a total of 8 weeks. Patients will visit the study center once weekly to receive their IV infusion of ofatumumab. To reduce the possibility of infusion reactions, the first dose of ofatumumab will be administered at a dose of 300 mg. If the initial 300 mg dose of ofatumumab is well tolerated, without occurrence of any infusion-associated AEs of ≥ grade 3, subsequent doses of ofatumumab (i.e., Week 2 through Week 8) will be at a dose of 2000 mg.

SUMMARY:
The risk of immunosuppression deters many patients from receiving fludarabine, while combination chemotherapy regimens are poorly tolerated by elderly or infirm chronic lymphocytic leukemia (CLL) patients. Previous studies by our group and others have shown that rituximab is safe and well tolerated when used as a single agent in patients with CLL. In addition, maintenance therapy with rituximab was well tolerated by CLL patients, with probable prolongation of progression-free survival (Hainsworth et al. 2003). Based on pre clinical and clinical studies indicating possible increased efficacy of ofatumumab in patients with CLL, we wish to develop an antibody-only regimen for older patients and patients who refuse fludarabine-based regimens.

ELIGIBILITY:
Inclusion Criteria:

1. CD20+ B-cell chronic lymphocytic leukemia (B-CLL) or small lymphocytic lymphoma according to NCI criteria (see Appendix B).
2. Previously untreated CLL or small lymphocytic lymphoma (SLL).
3. Patients must require treatment according to NCI-Working Group guidelines (see Appendix C).
4. Eastern Cooperative Oncology Group Performance Status (ECOG PS) of ≤2 (see Appendix A).
5. Laboratory values as follows ≤7 days of initiation of treatment:

   * Creatinine <3.0 mg/dL
   * Aspartate amino transferase (AST) or alanine amino transferase (ALT) and alkaline phosphatase (ALP) must be <3 x upper limit of normal (ULN)
   * Total bilirubin <1.5 x the institutional ULN
6. Patients must be hepatitis B sAg negative. Note: Patients who are HepB sAg negative but are HepB cAb positive (regardless of HepB sAb status) will NOT be allowed.
7. Women of childbearing potential must have a negative serum pregnancy test performed ≤7 days prior to start of treatment. Women of childbearing potential or men with partners of childbearing potential must use effective birth control measures during treatment. If a woman becomes pregnant or suspects she is pregnant while participating in this study, she must agree to inform her treating physician immediately.
8. Patients ≤ 65 years of age, or patients 18-64 years of age who have declined fludarabine-based regimens, are eligible.
9. Patient must be accessible for treatment and follow-up.
10. Patients must be able to understand the nature of this study, give written informed consent prior to study entry, and comply with study requirements.

Exclusion Criteria:

1. Previous therapy for CLL/SLL. (Patients who have received steroids or IVIG for autoimmune complications of CLL are eligible).
2. Current active hepatic or biliary disease (with the exception of patients with Gilbert's syndrome, asymptomatic gallstones, liver metastases, or stable chronic liver disease, per assessment by the treating physician).
3. Active bacterial or viral infection, or infection requiring intravenous antibiotic treatment at the time of accrual.
4. Central nervous system lymphoma/CLL.
5. Transformation of CLL to aggressive non-Hodgkin lymphoma (NHL) (i.e., Richters transformation).
6. History of other malignancy within 2 years of study entry which could affect compliance with the protocol or interpretation of results. Patients with a history of curatively treated basal or squamous cell carcinoma of the skin or in situ carcinoma of the cervix, low grade, early-stage, localized prostate cancer treated surgically with curative intent, ductal carcinoma in situ (DCIS) of the breast treated with curative intent, are generally eligible. These cases should be discussed with the study chair or study co-chair prior to enrollment.
7. Patients who are HepB sAg positive and/or HepB cAb positive.
8. Concurrent severe, intercurrent illness including, but not limited to, ongoing or active infection, or psychiatric illness/social situations that would limit compliance with study requirements.
9. Any condition that would prevent patient comprehension of the nature of, and risk associated with, the study.
10. A serious underlying medical condition that would impair the ability of the patient to receive protocol treatment.
11. A major surgical procedure, open biopsy, or significant traumatic injury ≤28 days of beginning treatment, or anticipation of the need for major surgery during the course of the study.
12. Treatment with any known non-marketed drug substance or experimental therapy within 5 terminal half lives or 4 weeks prior to visit 1, whichever is longer. Patients may not receive any other investigational or anti-cancer treatments while participating in this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 77 (Actual)
Dates: Start 2010-07; Primary Completion 2015-03 (Actual); Study Completion 2016-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ian Flinn, M.D., Study Chair — SCRI Development Innovations, LLC
Locations (13):
- United States (13):
  - Los Robles, Thousand Oaks, California
  - Florida Cancer Specialists, Fort Myers, Florida
  - Woodlands Medical Specialists, Pensacola, Florida
  - Northeast Georgia Medical Center, Gainesville, Georgia
  - Providence Medical Group, Terre Haute, Indiana
  - St. Louis Cancer Care, Chesterfield, Missouri
  - Portsmouth Regional Hospital, Portsmouth, New Hampshire
  - Hematology-Oncology Associates of Northern NJ, Morristown, New Jersey
  - Oncology Hematology Care, Cincinnati, Ohio
  - The Ohio State University, Columbus, Ohio
  - South Carolina Oncology Associates, Columbia, South Carolina
  - Chattanooga Oncology Hematology Associates, Chattanooga, Tennessee
  - Tennessee Oncology, Nashville, Tennessee

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg
Started | 33 | 44
Completed | 2 | 19
Not Completed | 31 | 25

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg | Total
Number analyzed (Participants) | 33 | 44 | 77
Age, Continuous [Median (Full Range); unit: years] | 75 [50 to 93] | 69 [47 to 88] | 72 [47 to 93]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 19 | 36
  Male | 16 | 25 | 41
Region of Enrollment [Number; unit: participants]
  United States | 33 | 44 | 77

OUTCOME MEASURES:

1. Secondary Outcome: Progression-free Survival (PFS)
Description: To assess the overall response rate of patients with previously untreated CLL or SLL receiving ofatumumab.
Time Frame: 18 months
Measure: Median (95% Confidence Interval); unit: months
Groups:
- Ofatumumab 1000mg: Ofatumumab 300mg IV Day 1 followed by ofatumumab 1000mg weekly for a total of 8 weeks
  Ofatumumab: IV infusion once weekly for a total of 8 weeks. Patients will visit the study center once weekly to receive their IV infusion of ofatumumab. To reduce the possibility of infusion reactions, the first dose of ofatumumab will be administered at a dose of 300 mg. If the initial 300 mg dose of ofatumumab is well tolerated, without occurrence of any infusion-associated AEs of ≥ grade 3, subsequent doses of ofatumumab (i.e., Week 2 through Week 8) will be at a dose of 1000 mg.
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg
Number analyzed (Participants) | 33 | 44
months | 19.8 [9.7 to NA] — Upper bound of the 95% confidence interval cannot be calculated as there is an insufficient number of events for this caluclation | 32.5 [26.6 to NA] — Upper bound of the 95% confidence interval cannot be calculated as there is an insufficient number of events for this caluclation

2. Primary Outcome: Overall Response Rate (ORR)
Description: The Number of Patients Who Experience an Objective Benefit From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR.
Time Frame: 18 months
Population: All patients who were evaluable for a response assessment
Measure: Number; unit: participants
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg
Number analyzed (Participants) | 28 | 44
participants | 15 | 30

3. Secondary Outcome: Number of Complete Responses
Description: The Number of Patients Who Experience a Complete Response From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Complete Response (CR), Disappearance of all target lesions
Time Frame: 18 Months
Population: All patients who were evaluable for a response assessment
Measure: Number; unit: participants
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg
Number analyzed (Participants) | 28 | 44
participants | 2 | 0

4. Secondary Outcome: Number of Partial Responses
Description: The Number of Patients Who Experience a Partial Response From Treatment. Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI or CT: Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions
Time Frame: 18 Months
Population: All patients who were evaluable for a response assessment
Measure: Number; unit: participants
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg
Number analyzed (Participants) | 28 | 44
participants | 13 | 30

5. Secondary Outcome: Safety of the Treatment Regimen
Description: Listing of all non-serious Adverse Events ocurring in 5% of patients or more
Time Frame: 18 Months
Measure: Number; unit: participants
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg
Number analyzed (Participants) | 33 | 44
participants
  Fatigue | 12 | 21
  Allergic reaction | 14 | 16
  Anemia | 14 | 13
  Pain | 9 | 14
  Platelet count decreased | 13 | 10
  Rash | 7 | 16
  White blood cell decreased | 10 | 9
  Cough | 5 | 13
  Diarrhea | 8 | 9
  Neutrophil count decreased | 7 | 10
  Dyspnea | 6 | 9
  Hyperglycemia | 4 | 11
  Edema | 8 | 6
  Nausea | 3 | 11
  Infections and infestations - Other, unspecified | 6 | 7
  Peripheral sensory neuropathy | 2 | 11
  Constipation | 2 | 10
  Insomnia | 3 | 9
  Psychiatric disorders - Other, unspecified | 5 | 7
  Arthralgia | 4 | 7
  Dizziness | 5 | 5
  Hyperhidrosis | 6 | 4
  Hypocalcemia | 4 | 5
  Aspartate aminotransferase increased | 6 | 2
  Blood bilirubin increased | 2 | 6
  Oral pain | 1 | 7
  Respiratory, thoracic and mediastinal disorders | 3 | 5
  Non-cardiac chest pain | 1 | 6
  Pruritus | 4 | 3
  Abdominal pain | 2 | 4
  Allergic rhinitis | 3 | 3
  Anorexia | 2 | 4
  Back pain | 2 | 4
  Fever | 2 | 4
  Gastrointestinal disorders - Other, unknown | 3 | 3
  Headache | 4 | 2
  Hypertension | 3 | 3
  Hyponatremia | 4 | 2
  Dysgeusia | 2 | 3
  Flushing | 1 | 4
  Gastroesophageal reflux disease | 3 | 2
  Hypoglycemia | 2 | 3
  Musculoskeletal and connective tissue disorders | 2 | 3
  Skin and subcutaneous tissue disorders - Other | 4 | 1
  Upper respiratory infection | 0 | 5
  Vomiting | 1 | 4
  Alanine aminotransferase increased | 2 | 2
  Blurred vision | 4 | 0
  Bruising | 1 | 3
  Chills | 1 | 3
  Creatinine increased | 1 | 3
  Hypokalemia | 1 | 3
  Infusion related reaction | 1 | 3
  Urinary frequency | 1 | 3
  Weight loss | 2 | 2

ADVERSE EVENTS:
Time Frame: 18 Months
Arm/Group | Ofatumumab 1000mg | Ofatumumab 2000mg
Serious Adverse Events (participants affected / at risk) | 3/33 | 2/44
Other Adverse Events (participants affected / at risk) | 32/33 | 42/44
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 1000mg (N=33) | Ofatumumab 2000mg (N=44)
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Anemia (Blood and lymphatic system disorders) | 1 | 0
Cholesterol high (Investigations) | 1 | 0
Creatinine increased (Investigations) | 0 | 1
Dysgeusia (Nervous system disorders) | 1 | 0
Edema (General disorders) | 1 | 0
Fever (General disorders) | 1 | 0
Gastrointestinal disorders - Other, hernia (Gastrointestinal disorders) | 1 | 0
Gastrointestinal disorders - Other, unknown (Gastrointestinal disorders) | 1 | 0
Hypoalbuminemia (Metabolism and nutrition disorders) | 1 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ofatumumab 1000mg (N=33) | Ofatumumab 2000mg (N=44)
Fatigue (General disorders) | 12 | 21
Allergic reaction (Immune system disorders) | 14 | 16
Anemia (Blood and lymphatic system disorders) | 14 | 13
Pain (General disorders) | 9 | 14
Platelet count decreased (Investigations) | 13 | 10
Rash (Skin and subcutaneous tissue disorders) | 7 | 16
White blood cell decreased (Investigations) | 10 | 9
Cough (Respiratory, thoracic and mediastinal disorders) | 5 | 13
Diarrhea (Gastrointestinal disorders) | 8 | 9
Neutrophil count decreased (Investigations) | 7 | 10
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 6 | 9
Hyperglycemia (Metabolism and nutrition disorders) | 4 | 11
Edema (General disorders) | 8 | 6
Nausea (Gastrointestinal disorders) | 3 | 11
Infections and infestations - Other, unspecified (Infections and infestations) | 6 | 7
Peripheral sensory neuropathy (Nervous system disorders) | 2 | 11
Constipation (Gastrointestinal disorders) | 2 | 10
Insomnia (Psychiatric disorders) | 3 | 9
Psychiatric disorders - Other, mood alteration (Psychiatric disorders) | 5 | 7
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 7
Dizziness (Nervous system disorders) | 5 | 5
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 6 | 4
Hypocalcemia (Metabolism and nutrition disorders) | 4 | 5
Aspartate aminotransferase increased (Investigations) | 6 | 2
Blood bilirubin increased (Investigations) | 2 | 6
Oral pain (Gastrointestinal disorders) | 1 | 7
Respiratory, thoracic and mediastinal disorders - Other, unknown (Respiratory, thoracic and mediastinal disorders) | 3 | 5
Non-cardiac chest pain (General disorders) | 1 | 6
Pruritus (Skin and subcutaneous tissue disorders) | 4 | 3
Abdominal pain (Gastrointestinal disorders) | 2 | 4
Allergic rhinitis (Respiratory, thoracic and mediastinal disorders) | 3 | 3
Anorexia (Metabolism and nutrition disorders) | 2 | 4
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 4
Fever (General disorders) | 2 | 4
Gastrointestinal disorders - Other, unknown (Gastrointestinal disorders) | 3 | 3
Headache (Nervous system disorders) | 4 | 2
Hypertension (Vascular disorders) | 3 | 3
Hyponatremia (Metabolism and nutrition disorders) | 4 | 2
Dysgeusia (Nervous system disorders) | 2 | 3
Flushing (Vascular disorders) | 1 | 4
Gastroesophageal reflux disease (Gastrointestinal disorders) | 3 | 2
Hypoglycemia (Metabolism and nutrition disorders) | 2 | 3
Musculoskeletal and connective tissue disorders - Other, unknown (Musculoskeletal and connective tissue disorders) | 2 | 3
Skin and subcutaneous tissue disorders - Other (Skin and subcutaneous tissue disorders) | 4 | 1
Upper respiratory infection (Infections and infestations) | 0 | 5
Vomiting (Gastrointestinal disorders) | 1 | 4
Alanine aminotransferase increased (Investigations) | 2 | 2
Blurred vision (Eye disorders) | 4 | 0
Bruising (Injury, poisoning and procedural complications) | 1 | 3
Chills (General disorders) | 1 | 3
Creatinine increased (Investigations) | 1 | 3
Hypokalemia (Metabolism and nutrition disorders) | 1 | 3
Infusion related reaction (General disorders) | 1 | 3
Urinary frequency (Renal and urinary disorders) | 1 | 3
Weight loss (Investigations) | 2 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor can review/embargo results communications prior to public release for a period that is >60 but =180 days from date submitted to sponsor, who may require changes to the communication in order to remove specifically identified confidential information (other than study data) and/or delay the proposed publication to enable the sponsor to seek patent protection for inventions. The PI may not publish its results until 18 mos. after the trial has been completed at all sites